CLINICAL TRIAL: NCT05727943
Title: Add-on Clioquinol in Drug-resistant Childhood Epilepsy: an Exploratory Study
Acronym: CLIOKID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Lieven Lagae, Principal Investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S 64647
Record Dates: First submitted 2022-12-23; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Epilepsy Intractable
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Clioquinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- add - on clioquinol (Experimental): Add-on clioquinol to concomitant anti seizure medications.
  Clioquinol - magistral suspension preparation (100mg/ml) - oral intake Exposure 2 weeks to low dose: 1 mg/kg/day Exposure 6 weeks to higher dose: 4 mg/kg/day
  Interventions: Drug: Clioquinol

INTERVENTIONS:
Drug: Clioquinol — add on clioquinol to concomitant ASM

SUMMARY:
In this exploratory trial, the potential anti-seizure activity of clioquinol in a small cohort of adolescents with drug-resistant epilepsy will be examined. Subjects will be exposed to clioquinol add-on for a period of maximum 8 weeks (2 weeks low dose, 6 weeks higher dose). The main hypothesis of the study is that 30% of the included subjects will be responders and that the median seizure frequency reduction will be at least 30%.

DETAILED DESCRIPTION:
In this exploratory phase 2 trial, adolescents with DRE will be exposed to clioquinol add-on for a period of maximum 8 weeks (2 weeks low dose, 6 weeks higher dose). During the trial concomitant anti-epileptic medication will be kept stable, so that only the add-on effect of clioquinol will be assessed. During a prospective baseline of 2 weeks, the number of seizures will be counted. The effect of first low dose (1mg/kg/day) and later higher dose (4mg/kg/day) of clioquinol on seizure frequency will be calculated using the typical epilepsy trial outcome measures: percent reduction of seizure frequency and number of patients with a >50% seizure frequency reduction ('responders').

PK samples will be collected in the first 4 patients pre-dose and 2, 4 and 8 hours post-dose, both at initiation of the lower dose (1mg/kg/day) and the higher dose (4mg/kg/day) and on visit 4. The obtained PK data will be compared with the available literature data. Since we cannot define 'absolute' PK values (yet), we use a relative stopping rule in this first phase. If >1 of the first 4 patients show a PK pattern which is more than 50% different (max PK values 50% above literature max values), the study will be ended in these 4 patients. If the dosages need to be changed for the following patients, a protocol amendment will be provided to the FAGG and the EC. In the following subjects, a simplified PK study will be done at both dosages to examine whether they follow the findings in the 4 exploratory patients. Here also, a stopping rule when the PK data is more than 50% higher than the PK data obtained in the first 4 patients will be used.

Not only the effect of the drug on seizure frequency will be calculated, but also the effect on seizure severity, overall impact of seizures, medication side effects, comorbidities, and overall QoL, using standardized questionnaires (NHS3 and PIES) (1, 2).

The main hypothesis of the study is that 30% of the included patients will be responders and that the median seizure frequency reduction will be at least 30%. These numbers are based on very similar trial results with new anti-epileptic drugs in drug-resistant childhood epilepsy.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this Trial must meet all of the following criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. In females with child bearing potential: negative pregnancy test or use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some intra-uterine devices, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomized partner
3. Age ≥ 12 years and < 18 years at time of inclusion
4. Weight ≥ 20 kg at time of inclusion
5. Well defined epilepsy history with convulsive seizures (with observable and countable motor component)
6. Drug-resistant epilepsy: before inclusion failure of at least 2 AEDs
7. Drug-resistant epilepsy: ≥ 4 seizures in the 2 week prospective period (baseline) before visit 2, not all (4) seizures observed in 1 of the 2 weeks. Baseline period can be extended with 1 or 2 weeks.
8. The patient is at the moment of inclusion on max 3 anti-epileptic drugs (VNS and ketogenic diet not included)

Exclusion Criteria:

1. Participant has a history of liver or kidney disease. Children with a co-existing active neuropathy (such as neuritis optica, transverse myelitis)
2. Asian ethnicity
3. Abnormal low blood level of vitamin B12 or Zn
4. Patients with hypothyroidism
5. Any disorder, which in the Investigator's opinion might jeopardize the participant's safety or compliance with the protocol
6. Any prior or concomitant treatment(s) that might jeopardize the participant's safety or that would compromise the integrity of the Trial
7. Exposure to clioquinol before the trial
8. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive
9. Participation in an interventional Trial with an IMP or device

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Responder rate : seizure frequency reduction | 8 weeks intervention
  Percentage of 50% responders after 2 weeks and 6 weeks exposure to low (1mg/kg/day) and higher doses (4mg/kg/day) of clioquinol respectively

SECONDARY OUTCOMES:
safety and Quality of Life assessment | 8 weeks intervention
  Safety during trial (systematic recording of adverse events)
  .

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Lagae, MD PhD, Principal Investigator — University Hospitals, University of Leuven
Locations (1):
- University Hospitals UZ Leuven, Leuven, Belgium